CLINICAL TRIAL: NCT03825406
Title: Prevalence of Wildtype Amyloid Among TAVR Patients With Impaired Hemodynamics
Brief Title: Prevalence of Wildtype Amyloid After TAVR
Status: Withdrawn | Type: Observational
Why Stopped: Dr. Bavry is recruiting the same patients for a NIH trial.
Sponsor: North Florida Foundation for Research and Education (Other)
Responsible Party: Sponsor
Other Study IDs: #: 201802928
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Those with abnormal vital signs after TAVR need to be willing to obtain a bone scan to evaluate for wildtype amyloidosis. Positive bone scan findings will require evaluation for primary amyloidosis with blood and urine monoclonal immunoglobulin testing. Primary amyloidosis is a different type of disease which requires different treatment.

DETAILED DESCRIPTION:
This research is interested in determining how common wildtype amyloidosis is after transcatheter aortic valve replacement (TAVR). Amyloidosis is a condition characterized by abnormal protein which can accumulate and impair various organs, including the heart. Research suggests that amyloidosis might be common among TAVR patients, but it is a condition that is not routinely evaluated for. We suspect that wildtype amyloidosis may be especially common among patients with abnormal vital signs after their TAVR procedure.

ELIGIBILITY:
Inclusion Criteria

* Patients that underwent a TAVR procedure at the Malcolm Randall VA Medical Center.
* Implant of current generation TAVR (i.e. Sapien S3, Evolut R, or Evolut Pro).
* Willingness to obtain bone scintigraphy if evidence of impaired hemodynamics after valve deployment.
* Willingness to have blood drawn
* Willingness to complete SF12 quality of life KCCQ

Exclusion Criteria:

--Patient that do not qualify for a TAVR procedure as normal clinical care

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research is interested in determining how prevalent wildtype amyloidosis is after transcatheter aortic valve replacement (TAVR) patients with impaired hemodynamics. Amyloidosis is a condition characterized by abnormal protein which can accumulate and impair various organs, including the heart. Research suggests that amyloidosis might be common among TAVR patients, but this condition is not routinely evaluated for. We suspect that wildtype amyloidosis may be especially common among patients with abnormal vital signs after their TAVR procedure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Number of participants who die or have poor quality of life as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 1 to 2 years post TAVR
  Measurement tool is the Kansas City Cardiomyopathy Questionnaire (KCCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bavry, MD, Principal Investigator — ACC AHA

REFERENCES:
- Available data/document: Study Protocol — http://va.gov — Type Study Protocol To request an electronic copy send email to Anthony.bavry@va.gov or debra.robertson1@va.gov
- Available data/document: Individual Participant Data Set — http://va.gov — De-identified data set for primary and secondary outcomes measures To request an electronic copy send email to Anthony.bavry@va.gov or Debra.robertson1@va.gov